CLINICAL TRIAL: NCT06819553
Title: Efficacy of Oral Potassium Citrate in Reducing Ureteral Stent Encrustation Post-Ureteroscopy
Brief Title: A Randomized Clinical Trial to Evaluate the Effectiveness of Oral Potassium Citrate in Preventing Ureteral Stent Encrustation in Patients Undergoing Ureteroscopy for Uric Acid Kidney Stones
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 571/13-Aug-2024
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-08

CONDITIONS: Urolithiasis; Stone Ureter
Keywords: stone disease; Oral Potassium Citrate
MeSH Terms: conditions — Urolithiasis; Ureterolithiasis | interventions — Potassium Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental Arm)Patients receiving potassium citrate. (Experimental): Oral potassium citrate (15 meq twice daily) to maintain urinary pH between 6.8 and 7.2.
  Interventions: Drug: Oral Potassium Citrate
- control arm (No Intervention): No oral potassium citrate or any other treatment for stent encrustation

INTERVENTIONS:
Drug: Oral Potassium Citrate — Evaluate the Effectiveness of Oral Potassium Citrate in Preventing Ureteral Stent Encrustation in Patients Undergoing Ureteroscopy for Uric Acid Kidney Stones
  Arms: Intervention Arm (Experimental Arm)Patients receiving potassium citrate.

SUMMARY:
This randomized clinical trial aims to evaluate the efficacy of oral potassium citrate in reducing ureteral stent encrustation following ureteroscopy for uric acid kidney stones. The study will assess whether potassium citrate, by raising urinary pH, can prevent encrustation on stents, potentially improving patient outcomes and reducing complications.

DETAILED DESCRIPTION:
Urolithiasis, particularly uric acid stones, is a prevalent condition with increasing incidence due to factors such as obesity and dietary habits. Ureteroscopy with stent placement is a common intervention for managing ureteral stones. However, the indwelling stents are prone to encrustation, which can lead to significant complications, including infection, obstruction, and discomfort for patients.

Potassium citrate, an alkalinizing agent, has been shown to prevent uric acid stone formation by raising urinary pH and dissolving existing stones. This trial aims to determine whether potassium citrate can also reduce encrustation on ureteric stents following ureteroscopy for uric acid stones.

In this prospective, randomized, controlled trial, patients undergoing ureteroscopy with stent placement for uric acid stones will be randomly assigned to either the intervention group (receiving potassium citrate) or a control group. The primary outcome is the rate of stent encrustation, which will be assessed using a modified scoring system after stent removal. Secondary outcomes include serum electrolyte levels, adverse events, and changes in urinary pH. All patients will be monitored regularly for changes in urine pH and adverse events during the study.

The findings from this trial may provide valuable insights into the role of potassium citrate in preventing ureteric stent encrustation, ultimately improving patient outcomes and reducing the need for additional interventions.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following criteria to be eligible)

* Age: ≥18 years old.
* Diagnosis: Patients undergoing ureteral stenting post-ureteroscopy for uric acid kidney stones.
* Urinary pH: ≤5.5 at baseline (acidic urine).
* Willingness to Participate: Patients who provide informed consent to participate in the study.

Exclusion Criteria (Participants will be excluded if they meet any of the following criteria) Renal Function: Patients with significantly impaired kidney function (elevated creatinine beyond normal limits).

Infections: History of febrile urinary tract infection (UTI) at the time of enrollment.

Metabolic Disorders:

Chronic kidney disease (CKD) Stage 3 or higher. History of hyperkalemia. Pregnancy: Pregnant or breastfeeding women. Residual Stones: Patients with residual stone burden after ureteroscopy that may confound outcomes.

Medication Interference: Patients on medications that significantly alter urinary pH (e.g., sodium bicarbonate, acetazolamide) or those contraindicated with potassium citrate.

Other Severe Comorbidities: Any condition that, in the investigator's judgment, would interfere with study participation or pose excessive risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
the rate of encrustation on the ureteral stents, which will be assessed after stent removal using a modified scoring system. | Stent removal, typically 4-6 weeks after ureteroscopy.
  The degree of encrustation on ureteral stents will be assessed using a modified encrustation scoring system upon stent removal. Encrustation severity will be categorized based on deposition on the stent surface, graded from no encrustation to severe encrustation.
  Stents will be examined macroscopically and, if applicable, under microscopy for calcium and uric acid deposits.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine - Zagazig University, Zagazig, Sharqia Province, Egypt